CLINICAL TRIAL: NCT03473860
Title: Study on the Relationship Between the Change of Total Cholesterol Content of Erythrocyte Membranes (CEM) and the Prognosis of Coronary Artery Disease in Real Clinical Practice
Brief Title: the Change of CEM and the Prognosis of Coronary Artery Disease in Real Clinical Practice
Acronym: CCEMPCAD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lu'an Municipal Hospital (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Sponsor
Other Study IDs: zjh2018315
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
Keywords: prognosis; all-cause mortality; myocardial infarction; stroke
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the change of total cholesterol content of erythrocyte membranes (CEM) in patients with coronary artery disease treated with secondary prevention drugs, and the correlation with the prognosis.

DETAILED DESCRIPTION:
In this clinical trial, plasma samples, the red cells and associated clinical data of patients with coronary artery disease were collected from Department of Cardiology of Lu'an Shili Hospital and the First Affiliated Hospital of Jinan University. Blood samples collected from all the participants at baseline (prior to the follow-up) and the time points of follow-up were placed into ordinary test tubes and stored at 4°C for less than 4 hours. After centrifuged, plasma and erythrocyte membranes was separated and stored at -80°C. The change of total cholesterol content of erythrocyte membranes (CEM) was measured. A follow-up form was designed according to the research purpose and discussed among the team members. The follow-up was performed through telephone by the trained investigators with good communication skills and knowledge on the diagnosis and treatment of coronary artery disease. Patients were followed up every six months from the day of discharge. The results of the follow-up were entered into the database, a process that was carried out by a designated person and double-checked by an independent person. The primary clinical endpoints were composite atherosclerotic cardiovascular disease outcomes, defined as nonfatal myocardial infarction, nonfatal stroke, or cardiovascular mortality. Secondary clinical endpoints were revascularization, including percutaneous coronary intervention and coronary artery bypass grafting, and Class IV heart failure requiring hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* First diagnosis of CAD through CAG;
* Aged 45-70.

Exclusion Criteria:

* Patients with severe liver or kidney damage;
* Taking statins within the last 3 months;
* Patients who had been diagnosed with CAD and treated with oral medication;
* Chronic diseases of the blood system;
* Familial hyperlipidemia patients;
* Patients combining autoimmune disease;
* Patients combining acute infectious disease;
* Patients who undertaken surgery or injury;
* Patients who combining cancer;
* Patients who taking glucocorticoid replacement therapy;
* Abnormal red blood cell (RBC) count (M: <4.0 or >5.5 × 1012/L; F: <3.5 or >5.0 × 1012/L) or abnormal hemoglobin (M: <120 or >160 g/L; F: <110 or >150 g/L).

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First diagnosis of CAD through CAG
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the change of CEM | before and 6-, 12-, 18-, 24- month after follow-up
  the change of CEM

SECONDARY OUTCOMES:
coronary revascularization | 24- months
  coronary revascularization
heart failure | 24- months
  heart failure
all-cause mortality | 24- months
  all-cause mortality
cardiovascular mortality | 24- months
  cardiovascular mortality
non-fatal myocardial infarction | 24- months
  non-fatal myocardial infarction
non-fatal stroke | 24- months
  non-fatal stroke